CLINICAL TRIAL: NCT04402294
Title: Individualized Closed Loop Transcranial Magnetic Stimulation (TMS) for Working Memory Enhancement
Brief Title: Individualized Closed Loop TMS for Working Memory Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Desmond Oathes, Dr., University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 832891; R01MH120811-05 (NIH)
Record Dates: First submitted 2020-05-04; First posted 2020-05-26 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Memory
Keywords: memory; healthy; TMS; MRI
MeSH Terms: interventions — Magnetic Resonance Imaging; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Task and resting fMRI will be used to determine an individualized brain target for each participant. In a subsequent session, participants will complete a task fMRI with repetitive TMS neuromodulation; during this session, various stimulation protocols will be interleaved with working memory task blocks to result in online brain readouts of the degree in which modulation affected the brain state in regards to working memory performance.
  Based on this testing, an optimal and sub-optimal TMS stimulation frequency will be determined for each individual participant. Each frequency will be administered separately across three stimulation days using a crossover design, with the order of frequencies being randomized and counterbalanced. Therefore, each subject will receive six days of TMS stimulation: three using the optimal frequency, and three using the sub-optimal frequency. The initial TMS/ task fMRI testing session will be completed at the midpoint and end of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Optimized TMS frequency, Then Sub-Optimal TMS Frequency (Experimental): In the first neuromodulation session, participants will receive rTMS using their optimal TMS frequency. After washout period of 1 week (minimum), the participants will start their second neuromodulation session using their sub-optimal TMS frequency instead.
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI); Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sub-Optimal TMS Frequency, Then Optimized TMS frequency (Experimental): In the first neuromodulation session, participants will receive rTMS using their sub-optimal TMS frequency. After washout period of 1 week (minimum), the participants will start their second neuromodulation session using their optimal TMS frequency instead.
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI); Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI) — Participants undergo resting-state and task-based fMRI to identify individualized transcranial magnetic stimulation (TMS) targets and determine optimal and sub-optimal stimulation frequencies. Additional fMRI scans are performed after each neuromodulation phase to assess changes following three days of stimulation at the optimal and sub-optimal frequencies.
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Participants first receive multiple rTMS frequencies during an fMRI scan to assess brain responses and determine individualized optimal and sub-optimal stimulation frequencies. They then complete two neuromodulation intervention periods, receiving rTMS at the identified optimal and sub-optimal frequencies. Each frequency is administered over three consecutive days, with the order of conditions randomized and counterbalanced.

SUMMARY:
The study is investigating working memory brain states by using transcranial magnetic stimulation (TMS) in combination with functional magnetic resonance imaging (fMRI). The study uses a novel, individualized targeting approach for TMS based on each subject's individual multi-modal fMRI data. The individualized target will be stimulated in a TMS/ fMRI imaging session to investigate working memory states and optimal stimulation frequencies.

DETAILED DESCRIPTION:
Prior to any study visits, all subjects will be pre-screened through a REDCap online self-report screening REDCap. The study involves 11 study visits.

The first study visit will consist of a consenting and extended screening visit. All participants will have the opportunity to ask questions before signing the electronic consent form. We will complete a semi-structured clinical interview and will demonstrate TMS to ensure the participant is comfortable with all study procedures. This visit will be completed both remote and in-person.

The second study visit will involve a 1-hour MRI scan. During the scan, the participant will complete multiple computerized tasks. The MRI scan will include both structural and functional scans, and those scans will be used to localize the stimulation target for the subsequent sessions.

The third study visit will be a 2-hour TMS/fMRI session, and the participant will engage in behavioral tasks while interleaved rTMS rounds are delivered at different excitatory frequencies (frequency range:

2Hz-20Hz). This scan will be used to determine the optimal stimulation frequency for the individual participant.

The fourth, fifth, and sixth study visits will involve neuromodulation with either the optimized frequency or the frequency least successful in moving a participants brain state, as determined from the third study visit. Each subject will receive ~3000 pulses in each session, including the pulses from the motor threshold determination. We will determine the stimulation amplitude by using the Stokes equation, which accounts for differences in cortical distance from the site relative to motor cortex (where the motor threshold is found).

The seventh study visit will involve a 1-hour TMS/fMRI session while the participant is engaging in a behavioral task. This visit is designed to examine brain and behavioral changes after the first round of neuromodulation.

The seventh and the eighth visit will be scheduled at least one week apart.

The eighth, ninth, and tenth study visits will mirror the fourth, fifth, and sixth study visits and will involve neuromodulation with either the optimized or least-optimized individual frequency. The order of optimized and least-optimized frequencies will be counterbalanced across participants between Visit 4-6 and Visit 8-10 (i.e., half of the participants will receive stimulations of the two frequencies in one order, and the other half will receive stimulations of the two frequencies in the reverse order). The eleventh visit will mirror the seventh visit and will examine brain and behavioral changes after the second round of neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

1)18-60 years old 2) Right handed 3) No psychiatric history as diagnosed by the SCID-V 4) Normal cognition 5) Capacity to give informed consent and follow study procedures 6) Sufficient command of English language to understand and respond to written as well as verbal instructions

Exclusion Criteria:

1. History of neurological disorder or traumatic brain injury (other than mild)
2. Unable to have an MRI scan, or current or prior medical condition that could interfere with the collection or interpretation of MRI data
3. Unable to receive TMS
4. Implanted devices, such as an aneurysm clip or cardiac pacemaker
5. History of stroke, epilepsy, or brain scarring
6. Recent use of psychoactive medications, as determined by investigators
7. Pregnant, nursing, or trying to become pregnant (self-attestation alone)
8. Color blindness
9. Otherwise determined by investigator to be unfit for study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 27 participants enrolled in the study, 2 withdrew before group assignment during the baseline MRI visit; one due to MRI-related discomfort and one due to scheduling conflicts.
Groups:
- Optimized TMS Frequency, Then Sub-Optimal TMS Frequency: In the first neuromodulation session, participants will receive rTMS using their optimal TMS frequency. After washout period of 1 week (minimum), the participants will start their second neuromodulation session using their sub-optimal TMS frequency instead.
  Repetitive Transcranial Magnetic Stimulation (rTMS): The investigators will create individualized TMS targets using deep learning methods on task and resting fMRI data to target working memory augmentation. The individualized target will be stimulated in a subsequent fMRI scan involving working memory task performance interleaved with repetitive TMS (rTMS) delivered at a variety of stimulation frequencies. Based on activation readouts in response to rTMS, an optimal and sub-optimal brain state frequency to impact working memory performance will be selected for each participant. Participants will receive rTMS at each frequency separately for three days (six days total), with the order of frequency randomly assigned and counterbalanced. Following each three day protocol, another fMRI working memory readout will be conducted to support the targeting and frequency selection algorithms.
- Sub-Optimal TMS Frequency, Then Optimized TMS Frequency: In the first neuromodulation session, participants will receive rTMS using their sub-optimal TMS frequency. After washout period of 1 week (minimum), the participants will start their second neuromodulation session using their optimal TMS frequency instead.
  Repetitive Transcranial Magnetic Stimulation (rTMS): The investigators will create individualized TMS targets using deep learning methods on task and resting fMRI data to target working memory augmentation. The individualized target will be stimulated in a subsequent fMRI scan involving working memory task performance interleaved with repetitive TMS (rTMS) delivered at a variety of stimulation frequencies. Based on activation readouts in response to rTMS, an optimal and sub-optimal brain state frequency to impact working memory performance will be selected for each participant. Participants will receive rTMS at each frequency separately for three days (six days total), with the order of frequency randomly assigned and counterbalanced. Following each three day protocol, another fMRI working memory readout will be conducted to support the targeting and frequency selection algorithms.
Period: Neuromodulation Week 1 (V4-V6)
Arm/Group | Optimized TMS Frequency, Then Sub-Optimal TMS Frequency | Sub-Optimal TMS Frequency, Then Optimized TMS Frequency
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: TMS/fMRI #2 (Visit 7)
Arm/Group | Optimized TMS Frequency, Then Sub-Optimal TMS Frequency | Sub-Optimal TMS Frequency, Then Optimized TMS Frequency
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Washout (at Least 7 Days)
Arm/Group | Optimized TMS Frequency, Then Sub-Optimal TMS Frequency | Sub-Optimal TMS Frequency, Then Optimized TMS Frequency
Started | 13 | 12
Completed | 12 | 11
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Insufficient study funds to continue with their participation. | 0 | 1
Period: Neuromodulation Week 2 (V8 - V10)
Arm/Group | Optimized TMS Frequency, Then Sub-Optimal TMS Frequency | Sub-Optimal TMS Frequency, Then Optimized TMS Frequency
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: TMS/fMRI #3 (Visit 11)
Arm/Group | Optimized TMS Frequency, Then Sub-Optimal TMS Frequency | Sub-Optimal TMS Frequency, Then Optimized TMS Frequency
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimized TMS Frequency, Then Sub-Optimal TMS Frequency | Sub-Optimal TMS Frequency, Then Optimized TMS Frequency | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.51 (5.98) | 22.67 (3.91) | 25.43 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time Changes During N-Back Task in Responses to Different TMS Frequencies
Description: During the TMS/fMRI scan, participants perform a working memory task (N-back). To evaluate how different repetitive TMS frequencies (5, 10, and 20 Hz) impact reaction time during N-back task, each rTMS train is followed by a block of the N-back task. A decoder identifies one frequency as optimal frequency and another as suboptimal frequency. Reaction Time during optimal, suboptimal, and no stimulation condition is assessed by taking average of reaction time on accurate trials with faster reaction times indicating better performance.
Time Frame: Single visit (~2 hours)
Population: All 19 participants underwent three different stimulation periods including Optimal, Suboptimal, and No Stimulation. Four subjects who completed the study were not included in the analysis due to technical issues leading to unreliable or missing data.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- N-Back Performance During Optimal Stimulation: Participants underwent optimal stimulation followed by the N-back task to assess its impact on performance. Accuracy and reaction time were used as performance metrics, with higher accuracy and/or faster responses indicating better performance.
- N-back Performance During Suboptimal Stimulation: Participants underwent suboptimal stimulation followed by the N-back task to assess its impact on performance. Accuracy and reaction time were used as performance metrics, with higher accuracy and/or faster responses indicating better performance.
- N-back Performance During No Stimulation: Participants also underwent periods of No Stimulation followed by the N-back task to assess its impact on performance. Accuracy and reaction time were used as performance metrics, with higher accuracy and/or faster responses indicating better performance.
Arm/Group | N-Back Performance During Optimal Stimulation | N-back Performance During Suboptimal Stimulation | N-back Performance During No Stimulation
Number analyzed (Participants) | 19 | 19 | 19
Seconds | 0.5853 (0.0980) | 0.5978 (0.1496) | 0.6012 (0.0961)
Statistical Analysis 1: Comparison: N-Back Performance During Optimal Stimulation vs N-back Performance During Suboptimal Stimulation vs N-back Performance During No Stimulation; ANOVA (Optimal vs Suboptimal vs No Stimulation); Test type: Other — Parametric inferential statistical test; p = 0.50, ANOVA — The threshold for statistical significance was set to p = 0.05; Group mean difference = 0.71

2. Primary Outcome: Accuracy Changes During N-Back Task in Responses to Different TMS Frequencies
Description: During the TMS/fMRI scan, participants perform a working memory task (N-back). To evaluate how different repetitive TMS frequencies (5, 10, and 20 Hz) impact accuracy during N-back task, each rTMS train is followed by a block of the N-back task. A decoder identifies one frequency as optimal frequency and another as suboptimal frequency. Accuracy during optimal, suboptimal, and no stimulation condition is assessed by taking average of all the trials with better accuracy indicating better performance.
Time Frame: Single visit (~2 hours)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | N-Back Performance During Optimal Stimulation | N-back Performance During Suboptimal Stimulation | N-back Performance During No Stimulation
Number analyzed (Participants) | 19 | 19 | 19
Percentage | 91.27 (16.30) | 90.71 (12.87) | 90.54 (13.14)
Statistical Analysis 1: Comparison: N-Back Performance During Optimal Stimulation vs N-back Performance During Suboptimal Stimulation vs N-back Performance During No Stimulation; ANOVA (Optimal vs Suboptimal vs No Stimulation); Test type: Other — Parametric inferential statistical test; p = 0.975, ANOVA — The threshold for statistical significance was set to p = 0.05; Group mean difference = 0.03

3. Primary Outcome: Reaction Time Changes in the Delayed Matching to Sample Task Following Optimal vs. Suboptimal rTMS Stimulation
Description: Each subject completes two 3-day neuromodulation sessions, one using their 'optimal' rTMS frequency, and the other using their 'suboptimal' rTMS frequency, as determined by their TMS/fMRI visit. After each neuromodulation session, subjects complete a working memory task (Delayed Match to Sample). The delay period reflects how long participants can retain the information in working memory. Common delay periods used in research, including our study, are 0 seconds, 4 seconds, and 12 seconds.The outcome measure shows the reaction time for each of these variables.
Time Frame: Up to 1 month
Population: Participants underwent three consecutive optimal and three consecutive suboptimal neuromodulation sessions in a randomized sequence. The optimal and suboptimal sessions were separated by at least one week to allow the effects of the stimulation to dissipate. the DMTS task consisted of three conditions including 0 sec, 4 sec, and 12 sec delay conditions. Four subjects who completed the study were not included in the analysis due to technical issues leading to unreliable or missing data.
Measure: Mean (Standard Error); unit: Reaction Time (sec)
Groups:
- Optimal Neuromodulation Day-1: Participants underwent three consecutive optimal and three consecutive suboptimal neuromodulation sessions in a randomized sequence. The optimal and suboptimal sessions were separated by at least one week to allow the effects of the stimulation to dissipate. This is for Day-1 of Optimal Stimulation.
- Optimal Neuromodulation Day-2: Participants underwent three consecutive optimal and three consecutive suboptimal neuromodulation sessions in a randomized sequence. The optimal and suboptimal sessions were separated by at least one week to allow the effects of the stimulation to dissipate. This is for Day-2 of Optimal Stimulation.
- Optimal Neuromodulation Day-3: Participants underwent three consecutive optimal and three consecutive suboptimal neuromodulation sessions in a randomized sequence. The optimal and suboptimal sessions were separated by at least one week to allow the effects of the stimulation to dissipate. This is for Day-3 of Optimal Stimulation.
- Suboptimal Neuromodulation Day-1: Participants underwent three consecutive optimal and three consecutive suboptimal neuromodulation sessions in a randomized sequence. The optimal and suboptimal sessions were separated by at least one week to allow the effects of the stimulation to dissipate. This is for Day-1 of Suboptimal Stimulation.
- Suboptimal Neuromodulation Day-2: Participants underwent three consecutive optimal and three consecutive suboptimal neuromodulation sessions in a randomized sequence. The optimal and suboptimal sessions were separated by at least one week to allow the effects of the stimulation to dissipate. This is for Day-2 of Suboptimal Stimulation.
- Suboptimal Neuromodulation Day-3: Participants underwent three consecutive optimal and three consecutive suboptimal neuromodulation sessions in a randomized sequence. The optimal and suboptimal sessions were separated by at least one week to allow the effects of the stimulation to dissipate. This is for Day-3 of Suboptimal Stimulation.
Arm/Group | Optimal Neuromodulation Day-1 | Optimal Neuromodulation Day-2 | Optimal Neuromodulation Day-3 | Suboptimal Neuromodulation Day-1 | Suboptimal Neuromodulation Day-2 | Suboptimal Neuromodulation Day-3
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
Reaction Time (sec)
  Reaction Time (0 sec delay) | 2.0173 (0.1423) | 1.7568 (0.0890) | 1.9316 (0.1862) | 2.0608 (0.1542) | 1.9118 (0.1068) | 1.9139 (0.1163)
  Reaction Time (4 sec delay) | 2.6640 (0.1936) | 2.4269 (0.1537) | 2.1726 (0.1292) | 2.3907 (0.1615) | 2.3268 (0.1694) | 2.4788 (0.2135)
  Reaction Time (12 sec delay) | 2.7351 (0.1588) | 2.5593 (0.1995) | 2.4400 (0.1602) | 2.4901 (0.1377) | 2.5741 (0.2054) | 2.6478 (0.2501)
Statistical Analysis 1: Comparison: Optimal Neuromodulation Day-1 vs Optimal Neuromodulation Day-2 vs Optimal Neuromodulation Day-3 vs Suboptimal Neuromodulation Day-1 vs Suboptimal Neuromodulation Day-2 vs Suboptimal Neuromodulation Day-3; ANOVA, with neuromodulation stimulation type (optimal vs. suboptimal), stimulation days (1 to 3), and delay (0, 4, or 12 seconds) as within-subject variables; Test type: Other — Parametric inferential statistical test; p = 0.097, ANOVA — The threshold for statistical significance was p = 0.05; Group mean difference = 2.05

4. Primary Outcome: Accuracy Changes in the Delayed Matching to Sample Task Following Optimal vs. Suboptimal rTMS Stimulation
Description: Each subject completes two 3-day neuromodulation sessions, one using their 'optimal' rTMS frequency, and the other using their 'suboptimal' rTMS frequency, as determined by their TMS/fMRI visit. After each neuromodulation session, subjects complete a working memory task (Delayed Match to Sample). The delay period reflects how long participants can retain the information in working memory. Common delay periods used in research, including our study, are 0 seconds, 4 seconds, and 12 seconds.The outcome measure shows the accuracy for each of these variables.
Time Frame: Up to 1 month
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Optimal Neuromodulation Day-1 | Optimal Neuromodulation Day-2 | Optimal Neuromodulation Day-3 | Suboptimal Neuromodulation Day-1 | Suboptimal Neuromodulation Day-2 | Suboptimal Neuromodulation Day-3
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
Percentage
  Accuracy (0 sec delay) | 84.2667 (3.2161) | 88.1011 (2.0073) | 83.9079 (3.6464) | 86.0638 (2.7408) | 87.8524 (2.3671) | 84.3748 (2.8921)
  Accuracy (4 sec delay) | 79.5037 (2.6388) | 78.1085 (2.7024) | 84.4127 (2.8358) | 78.2541 (3.0680) | 81.3003 (3.5756) | 77.5741 (2.8761)
  Accuracy (12 sec delay) | 79.4809 (2.7578) | 77.6172 (3.0897) | 88.0465 (2.5656) | 76.4133 (3.4818) | 76.1351 (3.1626) | 79.9014 (3.4101)
Statistical Analysis 1: Comparison: Optimal Neuromodulation Day-1 vs Optimal Neuromodulation Day-2 vs Optimal Neuromodulation Day-3 vs Suboptimal Neuromodulation Day-1 vs Suboptimal Neuromodulation Day-2 vs Suboptimal Neuromodulation Day-3; [analysis description as in outcome 3, analysis 1]; Test type: Other — Parametric Inferential Statistical Test; p = 0.644, ANOVA — The threshold for statistical significance was 0.05; Group mean difference = 0.63

5. Secondary Outcome: Reaction Time Changes in the Reaction Time Index Task Following Optimal vs. Suboptimal rTMS Stimulation
Description: Each subject completes two 3-day neuromodulation sessions, one using their 'optimal' rTMS frequency, and the other using their 'suboptimal' rTMS frequency, as determined by their TMS/fMRI visit. After each neuromodulation session, subjects complete a reaction time index task that acted as a control task. The outcome measure shows the reaction time.
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Optimal Neuromodulation Day-1 | Optimal Neuromodulation Day-2 | Optimal Neuromodulation Day-3 | Suboptimal Neuromodulation Day-1 | Suboptimal Neuromodulation Day-2 | Suboptimal Neuromodulation Day-3
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
Seconds | 0.716 (0.072) | 0.722 (0.108) | 0.687 (0.085) | 0.736 (0.117) | 0.713 (0.102) | 0.693 (0.093)
Statistical Analysis 1: Comparison: Optimal Neuromodulation Day-1 vs Optimal Neuromodulation Day-2 vs Optimal Neuromodulation Day-3 vs Suboptimal Neuromodulation Day-1 vs Suboptimal Neuromodulation Day-2 vs Suboptimal Neuromodulation Day-3; ANOVA, with neuromodulation stimulation type (optimal vs. suboptimal), and stimulation days (1 to 3) as within-subject variables; Test type: Other — Parametric inferential statistical test; p = 0.439, ANOVA — The threshold for statistical significance was p = 0.05; Group mean difference = 0.84

6. Secondary Outcome: Movement Time Changes in the Reaction Time Index Task Following Optimal vs. Suboptimal rTMS Stimulation
Description: Each subject completes two 3-day neuromodulation sessions, one using their 'optimal' rTMS frequency, and the other using their 'suboptimal' rTMS frequency, as determined by their TMS/fMRI visit. After each neuromodulation session, subjects complete a reaction time index task that acted as a control task. The outcome measure shows the movement time.
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Optimal Neuromodulation Day-1 | Optimal Neuromodulation Day-2 | Optimal Neuromodulation Day-3 | Suboptimal Neuromodulation Day-1 | Suboptimal Neuromodulation Day-2 | Suboptimal Neuromodulation Day-3
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
seconds | 0.411 (0.049) | 0.417 (0.087) | 0.381 (0.072) | 0.411 (0.098) | 0.406 (0.074) | 0.395 (0.076)
Statistical Analysis 1: Comparison: Optimal Neuromodulation Day-1 vs Optimal Neuromodulation Day-2 vs Optimal Neuromodulation Day-3 vs Suboptimal Neuromodulation Day-1 vs Suboptimal Neuromodulation Day-2 vs Suboptimal Neuromodulation Day-3; Optimal Neuromodulation Day-1, Optimal Neuromodulation Day-2, Optimal Neuromodulation Day-3, Suboptimal Neuromodulation Day-1, Suboptimal Neuromodulation Day-2, Suboptimal Neuromodulation Day-3; Test type: Other — Parametric inferential statistical test; p = 0.563, ANOVA — The threshold for statistical significance was p = 0.05; Group mean difference = 0.59

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study enrollment until study completion (up to 8 weeks)
Groups:
- Optimal rTMS Frequency: Three consecutive days of rTMS using their individualized optimal TMS frequency.
- Sub-Optimal rTMS Frequency: Three consecutive days of rTMS using their individualized sub-optimal TMS frequency.
Arm/Group | Optimal rTMS Frequency | Sub-Optimal rTMS Frequency
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal rTMS Frequency (N=24) | Sub-Optimal rTMS Frequency (N=24)
Headache (Nervous system disorders) | 2 (4) | 0 (0)
Jaw and Facial Muscle Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Tear Formation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anxiety/Panic/Discomfort (Nervous system disorders) | 1 (1) | 1 (1) — Anxiety, panic, or discomfort from procedures completed at the MRI scanner.

LIMITATIONS AND CAVEATS:
Enrollment goals were not met due to delays caused by COVID-19. Of the 23 subjects who completed the study, data from only 19 were analyzed. Technical issues with the remaining 4 subjects resulted in uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04402294/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04402294/ICF_001.pdf